CLINICAL TRIAL: NCT03266627
Title: A Pilot Study in the Treatment of Refractory Adenovirus (ADV) Infection With Related Donor ADV Cytotoxic T-Lymphocytes (ADV-CTLs)in Children, Adolescents and Young Adult Recipients
Brief Title: Adenovirus-specific Cytotoxic T-lymphocytes for Refractory Adenovirus Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Medical College of Wisconsin (Other); Nationwide Children's Hospital (Other); Johns Hopkins University (Other); University of California, San Francisco (Other); University of Colorado, Denver (Other); Indiana University (Other); Washington University School of Medicine (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 579; FD006363 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Adenovirus; Primary Immune Deficiency Disorder
Keywords: adenovirus; primary immune deficiency disorder; cytotoxic t-lymphocytes
MeSH Terms: conditions — Adenoviridae Infections; Primary Immunodeficiency Diseases

STUDY DESIGN:
Intervention Model Description: All eligible patients will receive one dose of CTLs at the same dose. Patients who meet the criteria may need additional CTL doses up to 5 total.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- patients with adenoviral infection (Experimental): patients will receive CTL dose x 1 with 2.5 × 10(4) CD3/kg for matched related donor and 0.5 × 104 CD3/kg for mis-matched related donor. Patients who don't respond to the first infusion may receive up to a total 5 CTL infusions.
  Interventions: Drug: cytotoxic t-lymphocytes

INTERVENTIONS:
Drug: cytotoxic t-lymphocytes — adenovirus specific cytotoxic t-lymphocytes will be collected and manufactured from HLA matched related or HLA mis-matched related donors and administered to eligible patients with refractory adenovirus or PID.
  Other Names: viral specific CTLs

SUMMARY:
Related donor Adenovirus (ADV) specific cytotoxic T cells (CTLs) manufactured with the Miltenyi CliniMACS Prodigy Cytokine Capture System will be administered intravenously in in children, adolescents and young adults with refractory ADV infection post Allogeneic Hematopoietic Stem Cell Transplantation (AlloHSCT), with primary immunodeficiencies (PID) or post solid organ transplant.

Funding Source: FDA OOPD

ELIGIBILITY:
1. Patients with Adenovirus infections post allogeneic HSCT, with primary immunodeficiencies or post solid organ transplant with:

   * Increasing or persistent quantitative ADV RT-PCR DNA copies despite two weeks of appropriate anti-viral therapy and/or
   * clinical symptoms attributed to adenovirus, including pneumonitis, hemorrhagic cystitis, colitis, hepatitis AND/OR
   * Medical intolerance to anti-viral therapies including:

     * grade 2 renal insufficiency secondary to cidofovir Consent: Written informed consent given (by patient or legal representative) prior to any study-related procedures.

   Performance Status > 30% (Lansky < 16 yrs and Karnofsky > 16 yrs) Age: 0.1 to 79 years

   Females of childbearing potential with a negative urine pregnancy test
2. Donor Eligibility Related donor available with a T-cell response to the viral MACS® GMP PepTivator antigen(s) of adenovirus.

   a. Third Party Related Allogeneic Donor: If original donor is not available or does not have a T-cell response: third party allogeneic donor (family donor > 1 HLA A, B, DR match to recipient) with a T-cell response at least to the viral MACS® GMP PepTivator antigen(s) of adenovirus.

   AND Allogeneic donor disease screening is complete similar to hematopoietic stem cell donors (Appendix 1).

   AND Obtained informed consents by donor or donor legally authorized representative prior to donor collection.
3. Patient exclusion criteria:

A patient meeting any of the following criteria is not eligible for the present study:

. Patient with acute GVHD > grade 2 or extensive chronic GVHD at the time of CTL infusion Patient receiving steroids (>0.5 mg/kg prednisone equivalent) at the time of CTL infusion Patient treated with donor lymphocyte infusion (DLI) within 4 weeks prior to CTL infusion Patient with poor performance status determined by Karnofsky (patients >16 years) or Lansky (patients ≤16 years) score ≤30% Concomitant enrollment in another experimental clinical trial investigating the treatment of refractory adenovirus infection(s) Any medical condition which could compromise participation in the study according to the investigator's assessment Known HIV infection Female patient of childbearing age who is pregnant or breast-feeding or not willing to use an effective method of birth control during study treatment.

Known hypersensitivity to iron dextran Patients unwilling or unable to comply with the protocol or unable to give informed consent.

Known human anti-mouse antibodies

-

Ages: 1 Month to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12 weeks after each infusion
  Patients will be followed for adverse events following each infusion of ADV CTLs
Incidence of Response to Treatment (Efficacy) | 12 weeks after last infusion
  Patients will be followed for improvement in viral infection by monitoring ADV PCR weekly for response to treatment with CTLs

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College
Locations (10):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Nationwide Children's Hosptial, Columbus, Ohio
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided